CLINICAL TRIAL: NCT00274469
Title: A Randomized, Open-Label, Parallel-Group, Multicentre, Phase II Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX™) 500 mg With Anastrozole (ARIMIDEX™) 1 mg as First Line Hormonal Treatment for Postmenopausal Women With Hormone Receptor Positive Advanced Breast Cancer
Brief Title: A Clinical Trial to Compare Efficacy and Tolerability of Faslodex With Arimidex in Patients With Advanced Breast Cancer
Acronym: FIRST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6995C00006; FIRST
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Breast Cancer
Keywords: oncology; cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Fulvestrant; Anastrozole

ARMS (2):
- 1 (Experimental): Fulvestrant
  Interventions: Drug: fulvestrant
- 2 (Active Comparator): Anastrozole
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: fulvestrant — 500 mg intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 1
Drug: anastrozole — 1 mg oral tablet
  Other Names: Arimidex; ZD1033
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of Faslodex (fulvestrant) with Arimidex (anastrozole) in postmenopausal women with hormone receptor positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hormone receptor positive advanced breast cancer, postmenopausal women

Exclusion Criteria:

* Previous treatment for advanced breast cancer (previous treatment for early breast cancer is allowed).

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2006-02-06 (Actual); Primary Completion 2008-01-10 (Actual); Study Completion 2017-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (37):
- United States (5):
  - Research Site, Frederick, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Teaneck, New Jersey
  - Research Site, Austin, Texas
  - Research Site, Duncanville, Texas
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Goiânia
  - Research Site, Jaú
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (7):
  - Research Site, Blagoevgrad
  - Research Site, Plovdiv
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- Czechia (5):
  - Research Site, Brno
  - Research Site, Jičín
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- France (3):
  - Research Site, Nice
  - Research Site, Poitiers
  - Research Site, Saint-Cloud
- Italy (2):
  - Research Site, Napoli
  - Research Site, Sassari
- Poland (2):
  - Research Site, Krakow
  - Research Site, Olsztyn
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Lleida
  - Research Site, Pontevedra
- United Kingdom (3):
  - Research Site, Derby
  - Research Site, Dundee
  - Research Site, Edinburgh

REFERENCES:
- See also: CSR-D6995C00006.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=405&filename=CSR-D6995C00006.pdf
- See also: D6995C00006FIRSToverall_survivalRevisedCSP_4_10_December_2014_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=405&filename=D6995C00006FIRSToverall_survivalRevisedCSP_4_10_December_2014_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women presenting with advanced breast cancer who had either never received endocrine therapy for advanced disease or had not received endocrine therapy in the previous 12 months in the adjuvant setting were recruited between 6th Feb 2006 and 11th July 2007.
Pre-assignment Details: 28 of the 233 enrolled patients were not randomized to treatment groups for the following reasons - 20 patients were incorrectly enrolled (ie did not comply with inclusion / exclusion criteria), 1 died, 1 had an adverse event, 4 voluntarily discontinued, 2 patients were not randomized for other non-specified reasons.
Groups:
- Fulvestrant 500 mg: Fulvestrant 500 mg
- Anastrozole 1 mg: Anastrozole 1 mg
Period: Overall Study
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Started | 102 (Number of patients randomized) | 103 (Number of patients randomized)
Completed | 23 (Number of patients ongoing study treatment at data cut-off) | 10 (Number of patients ongoing study treatment at data cut-off)
Not Completed | 79 | 93
Not completed — Death | 63 | 74
Not completed — Did not consent to OS follow-up | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (9.0) | 67.6 (9.3) | 67.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 103 | 205
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: A Clinical Benefit (CB) responder is defined as a patient having a best overall response of either complete response (CR), partial response (PR) or stable disease (SD) for at least 24 weeks evaluated according to modified RECIST. The Clinical Benefit Rate is the percentage of patients with CB.
Time Frame: From randomisation to data cut off (DCO) for primary analysis. The first and the last patients were enrolled on 6 Feb 2006 and 11 Jul 2007 respectively. The DCO for primary analysis was on 10th Jan 2008, 6 months after the last patient was enrolled.
Population: Full Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 102 | 103
Percentage of Participants | 72.5 | 67.0
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Non-Inferiority — Study is powered basing on 20% deficiency in benefit rate for Fulvestrant compared to Anastrozole; p = 0.386, Regression, Logistic — Null hypothesis: Fulvestrant has no difference with Anastrozole; Odds Ratio (OR) = 1.302, 95% CI 2-sided [0.717 to 2.380] — OR>1 favours Fulvestrant

2. Secondary Outcome: Objective Response Rate
Description: For each patient with measurable disease at baseline, the determination of the overall response for each visit was carried out using a SAS program per Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete Response (CR): Disappearance of all target lesion (TL) and non-target lesions (NTLs) and no new lesions. Partial Response (PR): At least a 30% decrease in the sum of longest diameter of TLs (compared to baseline), no progression of NTLs and no new lesions. Objective response rate is defined as percentage of patients with either CR or PR.
Time Frame: as for outcome 1
Population: Evaluable For Response Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 89 | 93
Percentage of Participants | 36.0 | 35.5
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.947, Regression, Logistic; Odds Ratio (OR) = 1.021, 95% CI 2-sided [0.556 to 1.874] — OR>1 favours Fulvestrant

3. Secondary Outcome: Time to Progression
Description: Time from randomization until earlier of disease progression or death. Progression was defined according to RECIST: a patient is determined to have progressed if they have progression of target lesions, clear progression of existing non-target lesions, or the appearance of one or more new lesions. Progression of target lesions is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum of LD recorded. Kaplan-Meier estimates of median for each treatment are reported.
Time Frame: as for outcome 1
Population: Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 102 | 103
Day | NA [173 to NA] — Median and 75% quartile not calculable | 381 [168 to NA] — 75% quartile not calculable
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.0496, Log Rank; Hazard Ratio (HR) = 0.6266, 95% CI 2-sided [0.3929 to 0.9991] — HR<1 favours Fulvestrant

4. Secondary Outcome: Time to Treatment Failure
Description: Time from randomization to treatment discontinuation
Time Frame: From randomisation to data cut off (DCO) for 75% treatment failure. The first and the last patients were enrolled on 6 Feb 2006 and 11 Jul 2007. The DCO for 75% treatment failure was on 26 Mar 2010, 32 months after the last patient was enrolled.
Population: Full analysis set.
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 102 | 103
Day | 536 [166 to 1303] | 387 [169 to 838]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.05, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.54 to 1.00] — HR<1 favours Fulvestrant
Statistical Analysis 2: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.04, Regression, Cox; Cox regression analysis of TTTF controlling for baseline covariates; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.52 to 0.98] — HR<1 favours Fulvestrant

5. Secondary Outcome: Time to Progression (Investigator Assessed)
Description: Time from randomization to disease progression (investigator assessed) or death from any cause. Progression was defined by investigator opinion, as patients did not have formal RECIST visits in the follow-up period after the data cut off for the primary analysis of the study.
Time Frame: as for outcome 4
Population: Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 102 | 103
Day | 712 [173 to 1331] | 400 [168 to 908]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.47 to 0.92] — HR<1 favours Fulvestrant
Statistical Analysis 2: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.01, Regression, Cox; Cox regression analysis of TTP (investigator assessed) controlling for baseline covariates; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.46 to 0.90] — HR<1 favours Fulvestrant

6. Post Hoc Outcome: Overall Survival
Description: Time from randomization to death (any cause)
Time Frame: From randomization to data cut off (DCO) for 65% OS analysis. The first and the last patients were enrolled on 6 Feb 2006 and 11 Jul 2007 respectively. The DCO for 65% OS analysis was on 15 Jul 2014, 7 years after the last patient was enrolled.
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 102 | 103
Month | 54.1 [29.7 to NA] — 75% quartile not calculable | 48.4 [28.6 to 78.5]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.041, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.50 to 0.98]
Statistical Analysis 2: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority; p = 0.126, Regression, Cox; Cox regression analysis of OS controlling for baseline covariates; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.54 to 1.08] — HR<1 favours Fulvestrant

ADVERSE EVENTS:
Time Frame: Non-serious adverse events = randomisation upto the point of data cut off for the primary efficacy analysis. Serious adverse events = randomisation up to the point of data cut off for the 65% overall survival analysis.
Description: First patient was enrolled on 6th Feb 2006. Non-serious AEs are reported from randomisation up to the data cut-off (DCO 10th Jan 2008) for the primary analysis (56 days after last injection and 30 days after last tablet). Serious AEs are reported from randomisation up to DCO for the 65% OS (15th July 2014).
  Note: All-Mortality is based on full population, while AEs and SAEs are based on safety population (1 less patient in Fulvestrant arm as it never received the randomised drug).
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
All-Cause Mortality (participants affected / at risk) | 63/102 | 74/103
Serious Adverse Events (participants affected / at risk) | 24/101 | 22/103
Other Adverse Events (participants affected / at risk) | 71/101 | 70/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500 mg (N=101) | Anastrozole 1 mg (N=103)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (2) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LACRIMAL DISORDER (Eye disorders) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (2)
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 0 (0) | 1 (1)
BLINDNESS (Eye disorders) | 1 (1) | 0 (0)
ANAL HAEMRROHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 2 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (3) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CANCERMETASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO THORAX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR HAEMORRAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500 mg (N=101) | Anastrozole 1 mg (N=103)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (14) | 8 (8)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 14 (19) | 10 (23)
CONSTIPATION (Gastrointestinal disorders) | 10 (12) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (9)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 7 (7)
DIZZINESS (Nervous system disorders) | 4 (4) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
FATIGUE (General disorders) | 1 (1) | 8 (8)
HEADACHE (Nervous system disorders) | 4 (26) | 13 (16)
HOT FLUSH (Vascular disorders) | 8 (8) | 14 (15)
HYPERTENSION (Vascular disorders) | 6 (6) | 2 (5)
INFLUENZA (Infections and infestations) | 1 (1) | 6 (6)
INJECTION SITE PAIN (General disorders) | 6 (14) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (10)
NAUSEA (Gastrointestinal disorders) | 10 (10) | 7 (8)
VOMITING (Gastrointestinal disorders) | 8 (10) | 3 (4)
ASTHENIA (General disorders) | 8 (14) | 8 (9)
DYSPEPSIA (Gastrointestinal disorders) | 2 (3) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (4) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 2 (2)
HIATUS HERNIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 1 (1)
ANAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 2 (2)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRODUODENITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RETCHING (Gastrointestinal disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 4 (4)
PYREXIA (General disorders) | 2 (2) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 3 (3) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 1 (3) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (3) | 0 (0)
INJECTION SITE PRURITUS (General disorders) | 2 (3) | 0 (0)
APPLICATION SITE PAIN (General disorders) | 1 (2) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (2) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
INJECTION SITE NODULE (General disorders) | 1 (1) | 0 (0)
IRRITABILITY (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 2 (2)
LETHARGY (Nervous system disorders) | 2 (2) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 2 (2)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
DIABETIC NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 0 (0) | 1 (1)
PAROSMIA (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
VITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 1 (3)
BRONCHITIS (Infections and infestations) | 3 (3) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 3 (3)
CYSTITIS (Infections and infestations) | 3 (3) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 2 (2)
TONSILLITIS (Infections and infestations) | 1 (1) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 1 (1)
ACARIASIS (Infections and infestations) | 1 (1) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ALLERGIC SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 2 (2) | 0 (0)
HYPERAEMIA (Vascular disorders) | 2 (2) | 0 (0)
PHLEBITIS (Vascular disorders) | 1 (1) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SCAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUBCUTANEOUS NODULE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 4 (4)
ANXIETY (Psychiatric disorders) | 3 (3) | 2 (2)
INSOMNIA (Psychiatric disorders) | 2 (2) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 2 (2) | 0 (0)
CRYING (Psychiatric disorders) | 0 (0) | 1 (1)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 1 (1)
NEUROSIS (Psychiatric disorders) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 2 (2)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 2 (2)
BREAST HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSPAREUNIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
GENITAL DISCHARGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 2 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0)
ACCOMMODATION DISORDER (Eye disorders) | 0 (0) | 1 (1)
CONJUNCTIVAL DISORDER (Eye disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0)
ERYTHEMA OF EYELID (Eye disorders) | 1 (1) | 0 (0)
EXOPHTHALMOS (Eye disorders) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1)
EYELID PTOSIS (Eye disorders) | 1 (1) | 0 (0)
MYOPIA (Eye disorders) | 0 (0) | 1 (1)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 3 (4)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 2 (2)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 2 (2)
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 0 (0) | 2 (2)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER TENDERNESS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1 (1) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 2 (2)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One patient in the ITT population was randomized to Fulvestrant 500 but did not receive drug and was excluded from the safety population. Hence, the safety population for Fulvestrant contained 101 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less